CLINICAL TRIAL: NCT00395837
Title: Efficacy of Lifestyle Changes in Modifying Practical Markers of Wellness and Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Anthony's Health Care (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #S2004.004
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Last update posted 2006-11-03 (Estimated); Status verified 2006-11

CONDITIONS: Aging
Keywords: Aging; Wellness; Aerobic exercise; Prevention
MeSH Terms: interventions — Exercise

INTERVENTIONS:
Behavioral: Aerobic exercise

SUMMARY:
To assess the impact of lifestylel changes upon measures of wellness and aging, in particular weight change, fitness measures, and cognitive performance. The hypothesis was that aerobic exercise would improve mental performance and measures of fitness.

DETAILED DESCRIPTION:
A 10-week, randomized control study conducted in a wellness center in St. Petersburg, Florida. Adults age 21-65, exercising less than 3 days/week. 56 subjects were randomized to a control or an intervention group. Subjects followed a diet with >30 grams of fiber and <16 grams of saturated fat daily, and were taught to reach 70-85% of their maximum heart rate 5-6 days/week, and to perform strength training 3 days/week, plus were asked to participate in 10-20 minutes of stress management activities daily. The study was designed to determine body composition, maximal aerobic capacity (VO2 max), total cholesterol/high-density lipoprotein (TC/HDL), and cognition.

Specific aspects ofcognitive performance were noted to increase with increasing levels of aerobic activity, but not with strength training, dietary fiber change, or stress managment.

Having established that the treatment group would exercise at different levels of intensity, additional subjects were recruited, and the cognitive performance of no exercise, moderate aerobic exercise, and frequent aerobic exercise could be compared with specific domains of cognitive performance: memory, psychomotor speed, reaction time, attention, and cognitive flexibility. The St Anthony's Institutional Review Board approved this research project.

ELIGIBILITY:
Inclusion Criteria:

* able to exercise 5-6 days per week

Exclusion Criteria:

* Free of major medical conditions, unable to exercise aerobically 5-6 days per week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2004-09; Study Completion 2006-05

PRIMARY OUTCOMES:
Cognitive performance (memory, psychomotor speed, reaction time, attention, cognitive flexibility)

SECONDARY OUTCOMES:
Cholesterol profile
Weight change
Body fat change
Changes in fitness (strength, flexibility, VO2max)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Masley, Principal Investigator — Medical Director
Locations (1):
- Carillon Wellness Center, St. Petersburg, Florida, United States